CLINICAL TRIAL: NCT03610126
Title: Comparison of Efficacy of BASKA Laryngeal Mask Airway in Either Volume or Pressure Controlled Ventilation in Laparoscopic Cholecystectomy Comparative Clinical Trial
Brief Title: BASKA Laryngeal Mask Airway in Either Volume or Pressure Controlled Ventilation in Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Principal Investigator, Assiut University
Other Study IDs: IRB: 17300212
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Ventilation
Keywords: BASKA mask; controlled ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- volume controlled ventilation: after induction of anesthesia and insertion of BASKA laryngeal mask airway mechanical ventilation of patients will be maintained with volume controlled ventilation mode
  Interventions: Procedure: volume controlled ventilation
- pressure controlled ventilation: after induction of anesthesia and insertion of BASKA laryngeal mask airway and mechanical ventilation of patients will be maintained with pressure controlled ventilation mode
  Interventions: Procedure: pressure controlled ventilation

INTERVENTIONS:
Procedure: volume controlled ventilation — the patients will be ventilated by volume controlled ventilation after insertion of the BASKA laryngeal mask airway
  Other Names: volume controlled
  Groups: volume controlled ventilation
Procedure: pressure controlled ventilation — the patients will be ventilated by pressure controlled ventilation after insertion of the BASKA laryngeal mask airway
  Other Names: pressure controlled
  Groups: pressure controlled ventilation

SUMMARY:
this study will be undertaken to compare the efficacy of BASKA mask in volume controlled and pressure controlled ventilation in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is one of the most commonly performed surgical procedures and the laryngeal mask airway (LMA) is the most common supraglottic airway device used by the anesthesiologists to manage airway during general anesthesia. Use of LMA has some advantages when compared to endotracheal intubation, such as quick and ease of placement, a lesser requirement for neuromuscular blockade and a lower incidence of postoperative morbidity. However, the use of the LMA in laparoscopy is controversial, based on a concern about increased risk of regurgitation and pulmonary aspiration. The ability of these devices to provide optimal ventilation during laparoscopic procedures has been also questioned. The most important parameter to secure an adequate ventilation and oxygenation for the LMA under pneumoperitoneum condition is its seal pressure of airway The BASKA mask is a novel supraglottic airway device. It has many of the features of other supraglottic airways, These include; A non-inflatable cuff, that it is continuous with the central channel of the device. As the pressure increases with positive pressure ventilation, the cuff itself is 'inflated', this may improve the seal, reduce leak, and make ventilation more efficient

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective cholecystectomy laparoscopic surgery.
* Age: 18-60 years.
* ASA physical status: I-II.

Exclusion Criteria:

* Patient refusal.
* History of cardiac disease, psychological disorders, respiratory diseases including asthma, renal or hepatic failure.
* Patients who have high risk of regurgitation or aspiration based on history of gastro esophageal reflux, hiatus hernia, diabetes and gross obesity.
* Neck pathology.
* Patients who predicted difficult airway (based on a history of difficult airway, mouth opening was less than 2.5 cm, inter-incisor distance < 20 mm, cervical spine pathology, modified Mallampati class III/IV, or thyromental distance < 65 mm).
* Preoperative sore throat.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ASA I&II in the age range 18-60 years of both sexes and scheduled for elective laparoscopic cholecystectomy surgery
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | Intra-operative
  the oropharyngeal leak airway pressure will be used as a primary outcome to compare the efficacy of BASKA mask in volume controlled and pressure controlled ventilation in laparoscopic cholecystectomy and measuring leak pressure.

SECONDARY OUTCOMES:
End tidal carbon dioxide | Intraoperative
  End tidal carbon dioxide measurement to determine efficacy of ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assiut university hospitals
Locations (1):
- Assiut university hospitals, Asyut, Assiut Governorate, Egypt